CLINICAL TRIAL: NCT05811910
Title: Role of Genetic Polymorphisms in Drug Induced Neuropathy in Children With Acute Lymphoblastic Leukemia
Brief Title: Genetic Polymorphisms in Drug Induced Neuropathy in Children With ALL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: IRCCS Burlo Garofolo (Other)
Responsible Party: Sponsor
Other Study IDs: 58/22
Record Dates: First submitted 2023-03-31; First posted 2023-04-13 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-03

CONDITIONS: Acute Lymphocytic Leukemia
Keywords: Acute lymphoblastic leukemia; GWAS; Toxicities
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Therapeutic success in childhood ALL reaches an outstanding success that currently relies upon risk stratification of patients with appropriate modulation of chemotherapy intensity based on underlying blasts' biological and molecular characteristics, and depth of initial treatment response. ALL polychemotherapeutic approaches share similar therapeutic scheme, with more intensive and toxic earlier phases (about 6 months) followed by a prolonged immunosuppressive regimen for maintenance (about 18 months). Protocols comprise glucocorticoids, antimetabolites, asparaginase, alkylating agents, antimitotic drugs antibiotics and, in case of Philadelphia positive ALL, anti-tyrosine kinase inhibitors combined together at different dosages and timing according to the patient's class of risk. ALL chemotherapeutic agents can damage nearly all organs. Some adverse reactions are extensions of the drugs' desired pharmacological effects on bone marrow and affect almost all children. Other adverse effects occur unpredictably in a smaller fraction of patients who, for unknown reasons, are more susceptible. Concerns about chemotherapy-related toxicities generated a significant need of finding predictive markers for the a priori identification of at-risk patients. Pharmacogenomics markers can be useful tools in clinics for tailoring therapy intensity on patients' genetic profile and in basic research for better understanding mechanistic and regulatory pathways of the biological functions associated with ALL treatment toxicities. Several genome wide association studies explored the landscape of ALL treatment-associated toxicities, discovering the contribution of important variants. Among these, TPMT single nucleotide polymorphisms (SNPs) have a well-recognized role in thiopurine-induced myelotoxicity. SNP rs924607 (C>T) in the promoter region of the gene encoding for the centrosomal protein 72 (CEP72) was associated with increased risk and severity of vincristine-related peripheral neuropathy. The aim of this study is to perform a GWAS in ALL children to provide insight into genetic loci affecting the occurrence of severe (grade III-V) vincristine-related peripheral neuropathy during induction therapy in the AIEOP protocols.

DETAILED DESCRIPTION:
Acute lymphoblastic leukemia (ALL) is the most common haematological cancer in children. Therapeutic success in childhood ALL reaches an outstanding success (5-years survival of about 85-90%), that currently relies upon risk stratification of patients with appropriate modulation of chemotherapy intensity based on underlying blasts' biological and molecular characteristics, and depth of initial treatment response. Although with some difference, worldwide ALL polychemotherapeutic approaches share the same therapeutic scheme, with more intensive and toxic earlier phases (to induce and consolidate remission, about 6 months), followed by a prolonged immunosuppressive regimen for maintenance (about 18 months). In particular, protocols comprise mostly glucocorticoids, antimetabolites, asparaginase, alkylating agents, antimitotic drugs antibiotics and, in case of Philadelphia positive ALL, anti-tyrosine kinase inhibitors combined together at different dosages and timing according to the patient's class of risk. ALL chemotherapeutic agents can damage nearly all organs. Some adverse reactions such as the hematological toxicities and their consequences (such as infections) are extensions of the drugs' desired pharmacological effects on bone marrow, and affect almost all children. Other adverse effects occur unpredictably in a smaller fraction of patients who, for unknown reasons, are more susceptible. High dose antimetabolites and DNA damaging drugs may cause a direct injury in healthy proliferating tissues, resulting in mucositis (about 40% of ALL patients). Corticosteroids may cause bone toxicities (such as osteoporosis, 5-70%), endocrinopathies (such as insulin resistance, hyperglycemia and prediabetes, 10-20%) and central nervous system toxicities (10-15%). Vincristine treatment is associated to peripheral motor or sensory neuropathy development (5-15%).8 Methotrexate crystals can precipitate in kidneys, inducing nephrotoxicity (about 3%).9 Asparaginase can lead to hypersensitivity reactions (30-70%) and pancreatitis (2-18%). Additional acute toxicities such as venous thromboembolism are rarer but still might contribute to the incidence of treatment related deaths. Concerns about chemotherapy-related toxicities have generated a significant need of finding predictive markers for the a priori identification of at-risk patients. In particular, pharmacogenomics markers can be useful tools both in clinics for tailoring therapy intensity on patients' genetic profile and in basic research for better understanding the mechanistic and regulatory pathways of the biological functions associated with ALL treatment toxicities. Several genome wide association studies (GWAS) -performed mainly by US/Canadian Children's Oncology Group (COG) ALL protocols- had explored and investigated the landscape of ALL treatment-associated toxicities, discovering the contribution of important variants. Among these, TPMT single nucleotide polymorphisms (SNPs) have a well-recognized role in thiopurine-induced myelotoxicity ad genotype-based guidelines are already available. SNP rs924607 (C>T) in the promoter region of the gene encoding for the centrosomal protein 72 (CEP72) was found to be associated with increased risk and severity of vincristine-related peripheral neuropathy. To author's knowledge, this is the only variant whose clinical validation is currently ongoing in a perspective clinical trial (Saint Jude Children Research Hospital (SJCRH) Total Therapy XVII, NCT03117751). The aim of this study is to perform a GWAS in ALL children to provide insight into genetic loci affecting the occurrence of severe (grade III-V) vincristine-related peripheral neuropathy during induction therapy in the AIEOP protocols

ELIGIBILITY:
Inclusion Criteria:

* Age >=1 year and <18 years old
* Newly diagnosed acute lymphoblastic leukemia (ALL)
* No Ph+ (BCR/ABL or t(9;22)-positive) ALL
* More than 4 weeks since prior steroids
* Written informed consent

Exclusion Criteria:

* Secondary ALL
* Prior disease that would preclude treatment with chemotherapy
* Evidence of pregnancy or lactation period
* Participation in another clinical study

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children aged 1-17 years with ALL
Sampling Method: Non-Probability Sample
Enrollment: 290 (Estimated)
Dates: Start 2021-03-30 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
To identify genetic loci affecting the occurrence of severe (grade III-V) vincristine-related peripheral neuropathy during induction therapy in the AIEOP-BFM protocols | At the end of the 2 year study period
  Toxicities will be assessed by clinicians using the National Cancer Institute Common Terminology Criteria for Adverse Events and graded as mild (grade I), moderate (grade II), serious/disabling (grade III), life-threatening (grade IV) or lethal (grade V). DNA will be genotyped by the lnfinium Omni2.5 BeadChip (Illumina) for a total number of markers of -2000000 SNP

CONTACTS AND LOCATIONS:
Overall Officials: Marco Rabusin, MD, Study Director — IRCCS materno infantile Burlo Garofolo
Locations (1):
- IRCCS materno infantile Burlo Garofolo, Trieste, Friuli Venezia Giulia, Italy

IPD SHARING:
Plan to Share IPD: No